CLINICAL TRIAL: NCT07363343
Title: Nifedipine and Enalapril vs Nifedipine and Labetalol for the Treatment of Postpartum Hypertension Study (NEPHRON)
Brief Title: Nifedipine and Enalapril vs Nifedipine and Labetalol for the Treatment of Postpartum Hypertension Study
Acronym: NEPHRON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-918
Record Dates: First submitted 2025-12-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Postpartum Preeclampsia
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; Enalapril; Enalaprilat; Labetalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nifedipine and Enalapril (Experimental): Nifedipine 60mg by mouth every twelve hours plus Enalapril 5mg by mouth every twelve hours
  Interventions: Drug: Nifedipine and Enalapril
- Nifedipine and Labetalol (Active Comparator): Nifedipine 60mg by mouth every twelve hours plus Labetalol 200mg by mouth every twelve hours
  Interventions: Drug: Nifedipine and Labetalol

INTERVENTIONS:
Drug: Nifedipine and Enalapril — Nifedipine 60mg by mouth every twelve hours plus Enalapril 5mg by mouth every twelve hours
  Other Names: Procardia and Vasotec
  Arms: Nifedipine and Enalapril
Drug: Nifedipine and Labetalol — Nifedipine 60mg by mouth every twelve hours plus Labetalol 200mg by mouth every twelve hours
  Other Names: Procardia and Trandete
  Arms: Nifedipine and Labetalol

SUMMARY:
To determine if nifedipine and enalapril will have better blood pressure control in the postpartum setting compared to nifedipine and labetalol.

DETAILED DESCRIPTION:
The primary objective is to assess the efficacy of enalapril on hypertension as a second line agent compared to labetalol in the postpartum period. This is a pragmatic, unblinded, randomized trial of postnatal patients with hypertension who are on nifedipine postpartum and require a second oral agent. Patients will be evaluated for eligibility and consented when they require initiation of a single oral antihypertension agent, if they require IV antihypertensive therapy, or if they are on a single oral antihypertensive medication intrapartum. After consenting for the study, patients will be initiated on extended release nifedipine 30 mg daily as the primary drug for treatment and increased to a maximum dose of 60 mg twice daily prior to starting a second agent. Nifedipine was chosen as the universal first line agent due to its longevity and diuretic properties. Medication up titration and initiation of a second antihypertensive agent will occur at the discretion of the treatment team. Medication adjustments are recommended when the majority (>50%) of recorded blood pressures are greater than 140 mm Hg systolic or 90 mm Hg diastolic during a 24-hour time period. This threshold was chosen based on our knowledge that higher systolic blood pressures are associated with increased cardiovascular outcomes. Women requiring an additional medication for treatment of hypertension will be randomly assigned to receive enalapril 5 mg twice daily or labetalol 200 mg twice daily for concomitant therapy.

Blood pressures will be analyzed at 24 hours after initiation of a second oral agent, 3 days following hospital discharge, 2 weeks postpartum and 6 weeks postpartum. Need for IV antihypertensive agents and an additional third oral agent will be reviewed. As per standard of care, participants will be asked to monitor their blood pressure (BP) at home twice daily and keep their own blood pressure log to share with their outpatient provider. Patients are instructed to notify their outpatient provider of elevated blood pressure readings according to the Postpartum Hypertension Information Sheet that will be provided to all study participants.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18 years or older
* Clinical diagnosis of hypertensive disorder in pregnancy (gestational hypertension, chronic hypertension, preeclampsia with or without severe features)
* Taking Nifedipine 60 mg every 12 hours for blood pressure control
* Persistently elevated blood pressure at/above 140/90 mmHg in a 24-hour time period or have one or more severe range blood pressure at/above 160/110 mmHg requiring a second antihypertensive medication
* English speaking

Exclusion Criteria:

* Taking ≥2 antihypertensive agents during pregnancy
* Heart block
* Heart rate <60 or >120 beats per minute
* Heart failure
* Creatinine >1.5 mg/dL
* Renal artery stenosis
* Active connective tissue disease
* Cerebrovascular accident
* Failed treatment or contraindications to nifedipine, enalapril or labetalol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postnatal women
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite postpartum hypertension treatment failure within 6 weeks postpartum | 6-weeks postpartum
  The primary outcome is a binary composite outcome, defined as the occurrence of any one or more of the following events within 6 weeks postpartum: Prolonged hospitalization, Hospital readmission for hypertension, Persistence of hypertension beyond 14 days postpartum, Requirement for acute treatment of severe-range hypertension. Participants experiencing at least one component will be classified as having met the composite outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Malshe, M.D., Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No